CLINICAL TRIAL: NCT06035432
Title: Trueness and Precision of Digital Models Obtained From Different Open-access Software Programs
Brief Title: Accuracy of Digital Models Using Open-access Software Programs
Status: Completed | Type: Observational
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Other Study IDs: Digital Models 2023
Record Dates: First submitted 2023-04-26; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Accuracy of Digital Dental Model

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Open access software 1
  Interventions: Other: Bluesky software
- Open access software 2
  Interventions: Other: 3D slicer software
- Non open access paid software 1
  Interventions: Other: OnDemand software
- Non open access paid software 2
  Interventions: Other: Mimics software

INTERVENTIONS:
Other: Bluesky software — Dental stone casts will be scanned with a desktop scanner and then STL files will be exported. Virtual 3D surface models will be obtained by Bluesky software.
  Groups: Open access software 1
Other: 3D slicer software — Dental stone casts will be scanned with a desktop scanner and then STL files will be exported. Virtual 3D surface models will be obtained by 3D slicer software.
  Groups: Open access software 2
Other: OnDemand software — Dental stone casts will be scanned with a desktop scanner and then STL files will be exported. Virtual 3D surface models will be obtained by OnDemand software.
  Groups: Non open access paid software 1
Other: Mimics software — Dental stone casts will be scanned with a desktop scanner and then STL files will be exported. Virtual 3D surface models will be obtained by Mimics software.
  Groups: Non open access paid software 2

SUMMARY:
Background: Despite the clear drive toward digital model transformation, there are limitations to some paid software necessary for digital model production. The aim of the study is to compare the accuracy of open-access software against paid software regarding the segmentation process to produce a digital model. Four groups of software programs will be assessed regarding their accuracy in the segmentation process to produce a digital dental model. The reference models will be scanned by a desktop scanner and will be set as the gold standard. The same models will be scanned by the same CBCT machine. The obtained DICOM data will be converted into STL files by four different software programs.

ELIGIBILITY:
Inclusion Criteria:

* Complete records of patients (upper and lower).
* Intact models with complete anatomy.
* Complete permanent dentition

Exclusion Criteria:

* Broken or damaged stone models.
* Models of patients with orthodontic appliances or dental prosthesis

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who are young adults attending the Periodontology, Oral Medicine, Diagnosis and Oral Radiology Department, Faculty of Dentistry, Alexandria University.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Deviation in digital models measurments | through study completion, up to 3 months
  3D deviation analysis will be done between the digital models of each participant and the reference model by reverse engineering 3-Matics software (Materialise NV, Belgium, Version 11.0). Each two STL models will be imported into the software. The mean deviation difference (measured in mm) will be calculated by 'Analyse' tool present in the software

SECONDARY OUTCOMES:
Linear measurements | through study completion, up to 3 months
  Each digital model will be measured in the three dimensions:
  1. Anteroposterior (the canine cusp tip to the mesiobuccal cusp tip of the first molar on the right side).
  2. Transverse (inter-canine and inter-molar).
  3. Vertical (the canine height, which is measured from the cusp tip to the gingival margin of the right canine by a line parallel to the long axis of the tooth).
Teeth crown width | through study completion, up to 3 months
  For all teeth (twelve measurements for each arch), first molar to first molar, in both arches, the tooth measurements will include the mesiodistal widths from point contact to point contact.

CONTACTS AND LOCATIONS:
Overall Officials: Noha ElKersh, PhD, Principal Investigator — Alexandria University, Faculty of Dentistry
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt